CLINICAL TRIAL: NCT07090096
Title: A Randomized Controlled Trial of a Nutritional Intervention for Endometriosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sanjay Agarwal, MD, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 806685
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Endometriosis
Keywords: endometriosis, pain, quality of life, inflammatory markers, diet, nutrition
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled design with an active and control arms
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm which will receive the intervention (Experimental): This group will receive the dietary intervention
  Interventions: Other: A whole food plant based diet
- Control (No Intervention): This group with continue on their usual diet

INTERVENTIONS:
Other: A whole food plant based diet — A whole food plant based (WFPB) diet
  Other Names: WFPB
  Arms: Experimental arm which will receive the intervention

SUMMARY:
This randomized, controlled study will investigate the efficacy of a dietary intervention for women with endometriosis. Participants will be randomly assigned to follow a whole food plant-based (intervention) diet or stay on their usual (control) diet for 12 weeks.

DETAILED DESCRIPTION:
This randomized, controlled study will investigate the efficacy of a dietary intervention for women with endometriosis. Participants will be randomly assigned to follow a whole food plant-based (intervention) diet or stay on their usual (control) diet for 12 weeks. We want to see if this diet improves and pain and quality of life in women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study visits, procedures, requirements, and availability for the duration of the study
3. Women with a surgical, imaging, or clinical diagnosis of endometriosis
4. Age 18-45 years
5. Stable health condition and medications for the past 3 months
6. Modified Biberoglu and Behrman (B&B) pelvic pain score of at least 5/9
7. Willing to be randomly assigned to either an active or a control group
8. Agreement to adhere to Lifestyle Considerations throughout the study duration

Exclusion Criteria:

1. Smoking or drug abuse during the past six months
2. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
3. Already following a WFPB diet
4. Pregnant or breastfeeding, or plans of pregnancy within the study period
5. Hysterectomy or ovariectomy
6. Fibroids, ovarian cysts, pelvic inflammatory disease
7. Endocrine inflammatory conditions, such as Cushing's syndrome, Hashimoto's thyroiditis, Graves' disease, type 1 diabetes mellitus, and Addison's disease
8. Evidence of an eating disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Total pain score | 12 weeks
  Change in total VAS for dysmenorrhea, dyspareunia and non-menstrual pelvic pain

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay K Agarwal, MD, Principal Investigator — UCSD
Locations (1):
- UCSD Health, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No
It will be proprietary